CLINICAL TRIAL: NCT00145613
Title: Haploidentical Stem Cell Transplantation Utilizing T-Cell Depletion as Therapy for Patients With Refractory Hematological Malignancies
Brief Title: Haploidentical Stem Cell Transplant for Treatment Refractory Hematological Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Gregory Hale, M.D. / Principal Investigator, St. Jude Children's Research Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REFSCT
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-02

CONDITIONS: Acute Lymphoblastic Leukemia (ALL); Acute Myeloid Leukemia (AML); Secondary AML; Myelodysplastic Syndrome (MDS); Secondary MDS; Chronic Myeloid Leukemia; Juvenile Myelomonocytic Leukemia (JMML); Paroxysmal Nocturnal Hemoglobinuria (PNH); Lymphoma, Non-Hodgkin; Hodgkin Disease
Keywords: Haploidentical stem cell transplant; High risk hematologic malignancies; Allogeneic stem cell transplant; Mismatched family member stem cell donor
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myelomonocytic, Juvenile; Hemoglobinuria, Paroxysmal; Lymphoma, Non-Hodgkin; Hodgkin Disease | interventions — Stem Cell Transplantation; Antibodies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Procedure: Stem Cell Transplantation; Device: Miltenyi Biotec CliniMACS; Drug: Systemic chemotherapy and antibodies

INTERVENTIONS:
Procedure: Stem Cell Transplantation — An infusion of HLA mismatched family member donor stem cells processed through the use of the investigational Miltenyi Biotec CliniMACS device.
Device: Miltenyi Biotec CliniMACS — stem cell selection device
Drug: Systemic chemotherapy and antibodies — Transplant recipients received a non-TBI based reduced intensity conditioning regimen consisting of OKT-3, Fludarabine Thiotepa, and Melphalan. Rituximab was administered within 24 hours of the transplant in an effort to prevent PTLPD. In addition to T-cell depletion of the haploidentical stem cell product, Mycophenolate mofetil was provided as prophylaxis for GVHD.
  Other Names: Allogeneic stem cell transplant,; Mismatched family member donor stem cell transplant; Haploidentical donor stem cell transplant,; Reduced intensity conditioning regimen,; T-cell depletion donor stem cell processing

SUMMARY:
Relapsed disease is the most common cause of death in children with hematological malignancies. Patients who fail high-intensity conventional chemotherapeutic regimens or relapse after stem cell transplantation have a poor prognosis. Toxicity from multiple therapies and elevated leukemic/tumor burden usually make these patients ineligible for the aggressive chemotherapy regimens required for conventional stem cell transplantation. Alternative options are needed. One type of treatment being explored is called haploidentical transplant.

Conventional blood or bone marrow stem cell transplant involves destroying the patient's diseased marrow with radiation or chemotherapy. Healthy marrow from a donor is then infused into the patient where it migrates to the bone marrow space to begin generating new blood cells. The best type of donor is a sibling or unrelated donor with an identical immune system (HLA "match"). However, most patients do not have a matched sibling available and/or are unable to identify an acceptable unrelated donor through the registries in a timely manner. In addition, the aggressive treatment required to prepare the body for these types of transplants can be too toxic for these highly pretreated patients. Therefore doctors are investigating haploidentical transplant using stem cells from HLA partially matched family member donors.

Although haploidentical transplant has proven curative in many patients, this procedure has been hindered by significant complications, primarily regimen-related toxicity including graft versus host disease (GVHD), and infection due to delayed immune reconstitution. These can, in part, be due to certain white blood cells in the graft called T cells. GVHD happens when the donor T cells recognize the patient's (the host) body tissues are different and attack these cells. Although too many T cells increase the possibility of GVHD, too few may cause the recipient's immune system to reconstitute slowly or the graft to fail to grow, leaving the patient at high-risk for infection. However, the presence of T cells in the graft may offer a positive effect called graft versus malignancy or GVM. With GVM, the donor T cells recognize the patient's malignant cells as diseased and, in turn, attack these diseased cells.

For these reasons, a primary focus for researchers is to engineer the graft to provide a T cell depleted product to reduce the risk of GVHD, yet provide a sufficient number of cells to facilitate immune reconstitution, graft integrity and GVM.

In this study, patients were given a haploidentical graft engineered to with specific T cell parameter values using the CliniMACS system. A reduced intensity, preparative regimen was used to reduce regimen-related toxicity and mortality. The primary goal of this study is to evaluate overall survival in those who receive this study treatment.

DETAILED DESCRIPTION:
Secondary objectives for this protocol are to 1) assess the kinetics of lymphohematopoietic reconstitution and 2) describe the short and long-term (up to 5 years post- transplant) toxicity of haploidentical stem cell transplantation, including GVHD, in children with refractory hematological malignancies.

ELIGIBILITY:
Inclusion Criteria: Refractory hematological malignancies (chemoresistant relapse or primary induction failure) including:

* Acute lymphoblastic leukemia (ALL), must have isolated or combined bone marrow relapse or primary induction failure. Patients with extramedullary relapse are not eligible unless they have previously received a stem cell transplant
* Acute myeloid leukemia (AML) >25% blasts in bone marrow
* Secondary AML
* Myelodysplastic syndrome (MDS)
* Secondary MDS
* Chronic myeloid leukemia (CML)
* Juvenile myelomonocytic leukemia (JMML)
* Paroxysmal nocturnal hemoglobinuria (PNH)
* Non-Hodgkin's lymphoma (NHL)*
* Hodgkin's Disease (HD)*

  *Patients with lymphomas must have failed standard non-cross reactive combination salvage chemotherapy with or without radiation therapy followed by autologous stem cell transplant or patients with chemo resistant disease
* If patient has had previous stem cell transplant, must not be no earlier than 3 months from previous date of transplant
* Patients with shortening fraction greater than or equal to 25%
* Patients with creatinine clearance greater than or equal to 40cc/min/1.73m^2
* Patients with FVC greater than or equal to 40% of predicted, or pulse oximetry greater than or equal to 92% on room air
* Patients with a performance score (Lansky/Karnofsky) of greater than or equal to 50
* Must have a suitable family member donor that is HIV negative, greater than or equal to 18 years of age available for stem cell donation

Exclusion Criteria:

* Patients with a known allergy to murine products
* (Female Patients) Patient is pregnant
* Female Patients) Patient is lactating

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2003-06; Primary Completion 2006-07 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
To ask in terms of one-year survival the efficacy of haploidentical stem cell transplantation in children with refractory hematological malignancies. | July 2006

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Hale, M.D., Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org